CLINICAL TRIAL: NCT03793608
Title: A Study to Evaluate the Efficacy and Safety of Dupilumab Monotherapy in Pediatric Patients With Peanut Allergy
Brief Title: Study to Evaluate Dupilumab Monotherapy in Pediatric Patients With Peanut Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R668-ALG-1702; 2018-003133-15 (EudraCT Number)
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Results first posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dupilumab (Experimental): Open label weight base subcutaneous (SC) injection every two (Q2) weeks.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Dupilumab weight-based dosing will be administered subcutaneously (SC) in a single-use, pre-filled syringe every two weeks (Q2W)
  Other Names: REGN668; IL4R; Dupixent; SAR231893

SUMMARY:
The primary objective of the study is to assess the tolerability of peanut protein in pediatric patients (6-17 years old) treated with dupilumab monotherapy, in which tolerability is defined as the proportion of patients who safely pass a double-blind placebo-controlled food challenge (DBPCFC) at week 24.

The secondary objectives are:

* To determine whether dupilumab treatment improves peanut tolerability, defined as a change in the cumulative tolerated dose (log transformed) of peanut protein during a DBPCFC
* To evaluate the safety and tolerability of dupilumab treatment in peanut allergic patients
* To evaluate the effects of dupilumab treatment on the levels of peanut-specific Immunoglobulin E (IgE)
* To evaluate the treatment effect of dupilumab on the average wheal size after a titrated skin prick test (SPT), as measured by area under curve (AUC) of the average wheal size induced by peanut extract at different concentrations
* To assess the incidence of treatment-emergent anti-drug antibodies (ADA) to dupilumab in patients over time

ELIGIBILITY:
Key Inclusion Criteria:

* Patient has a clinical history of allergy to peanuts or peanut-containing foods (symptom[s] of reaction due to exposure).
* Experience dose-limiting symptoms at or before the challenge dose of peanut protein on screening DBPCFC conducted in accordance with Practical Issues in Allergology, Joint United States/European Union Initiative (PRACTALL) guidelines. And not experiencing dose limiting symptoms to placebo
* Serum IgE to peanut of ≥10 kilo units (kUA)/L and/or a SPT to peanut ≥8 mm compared to a negative control
* Patients/legal guardians must be trained on the proper use of the epinephrine autoinjector device to be allowed to enroll in the study
* Patients with other known food allergies must agree to eliminate these other food items from their diet so as not to confound the safety and efficacy data from the study

Key Exclusion Criteria:

* Any previous exposure to marketed dupilumab or dupilumab in a clinical trial
* Member of the clinical site study team or his/her immediate family
* History of other chronic disease (other than asthma, AD, or allergic rhinitis) requiring therapy
* History of frequent or recent severe, life-threatening episode of anaphylaxis or anaphylactic shock as defined by more than 3 episodes of anaphylaxis within the past year and/or an episode of anaphylaxis within 60 days of screening DBPCFC
* History of eosinophilic gastrointestinal disease
* History of eosinophilic granulomatosis with polyangiitis
* Severe, unstable asthma at time of enrollment or any patient with Forced Expiratory Volume in 1 Second (FEV1) <80% of predicted or asthma control questionnaire (ACQ)>1.5
* Use of systemic corticosteroids within 2 months prior to screening

Note: Other protocol Inclusion/Exclusion Criteria apply

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (9):
- United States (6):
  - Regeneron Investigational Site, Mountain View, California
  - Regeneron Investigational Site, Tampa, Florida
  - Regeneron Investigational Site, Indianapolis, Indiana
  - Regeneron Investigational Site, Ypsilanti, Michigan
  - Regeneron Investigational Site, Great Neck, New York
  - Regeneron Investigational Site, The Bronx, New York
- Canada (3):
  - Regeneron Investigational Site, Hamilton, Ontario
  - Regeneron Investigational Site, Toronto, Ontario
  - Regeneron Investigational Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual de-identified participant data will be made available once the indication has been approved by a regulatory body, if there is participant consent and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to study documents (including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan) that support the methods and findings reported in a manuscript. Individual de-identified participant data will be made available once the indication has been approved by a regulatory body, if there is participant consent and there is not a reasonable likelihood of participant re-identification.
URL: https://vivli.org/

REFERENCES:
- [Derived] Chinthrajah RS, Sindher SB, Nadeau KC, Leflein JG, Spergel JM, Petroni DH, Jones SM, Casale TB, Wang J, Carr WW, Shreffler WG, Wood RA, Wambre E, Liu J, Akinlade B, Atanasio A, Orengo JM, Hamilton JD, Kamal MA, Hooper AT, Patel K, Laws E, Mannent LP, Adelman DC, Ratnayake A, Radin AR. Dupilumab as an Adjunct to Oral Immunotherapy in Pediatric Patients With Peanut Allergy. Allergy. 2025 Mar;80(3):827-842. doi: 10.1111/all.16420. Epub 2024 Dec 14. PMID 39673367
- [Derived] Ghelli C, Costanzo G, Canonica GW, Heffler E, Paoletti G. New evidence in food allergies treatment. Curr Opin Allergy Clin Immunol. 2024 Aug 1;24(4):251-256. doi: 10.1097/ACI.0000000000000999. Epub 2024 May 30. PMID 38814736

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-five participants met eligibility criteria. One of the 25 participants was randomized under the original double-blind placebo-controlled protocol and received placebo-matching dupilumab. Following implementation of Protocol Amendment 1, 24 participants were enrolled under the open-label design & received open-label treatment with dupilumab.
Pre-assignment Details: A double-blind placebo-controlled food challenge (DBPCFC) consisting of increasing amounts of peanut protein up to a cumulative total of 144 mg and a matching placebo challenge consisting of placebo material (oat protein) were given to confirm current peanut allergy. Food challenges were performed on different days in random order (1-day placebo, 1-day peanut protein), at least 24 hours, but not more than 7 days, apart. Both food challenge days were required to evaluate eligibility.
Groups:
- Placebo: Participant enrolled under original double-blind protocol design randomized to receive placebo matched to dupilumab from Day 1 up to Week 22. At Week 24, all participants underwent a DBPCFC up to 2044 mg peanut protein (cumulative) or placebo to assess tolerability.
- Dupilumab: Participants enrolled under open-label treatment protocol with weight of greater than or equal to (>=) 20 kilograms (kg) and less than (<) 60 kg received a subcutaneous (SC) injection of dupilumab 200 mg every 2 weeks (Q2W) after a loading dose of 400 mg on Day 1 up to Week 22; participants with weight of >=60 kg received a SC injection of dupilumab 300 mg Q2W after a loading dose of 600 mg on Day 1 up to Week 22. At Week 24, all participants underwent a DBPCFC up to 2044 mg peanut protein (cumulative) or placebo to assess tolerability.
Period: Overall Study
Arm/Group | Placebo | Dupilumab
Started | 1 | 24
Treated | 1 | 24
Safety Analysis Set (SAF) (The safety analysis set (SAF) included all participants who received dupilumab. All efficacy and safety variables were analyzed using SAF.) | 0 (1 participant randomized to placebo was not analyzed and thus excluded from analyses.) | 24
Completed | 1 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: SAF(all participants who received dupilumab)
Arm/Group | Dupilumab
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.7 (3.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Treated With Dupilumab Who Passed a DBPCFC With at Least 444 mg (Cumulative) Peanut Protein at Week 24
Description: Symptoms considered to be allergic were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions. The scale is Grade 1 (Mild) through 5, the higher the grade, the more severe the allergic reaction. Participants were considered to have passed the DBPCFC if they did not experience any objective Grade 1 reaction. Percentage of participants treated with dupilumab who passed the DBPCFC with at least 444 mg (cumulative) peanut protein at Week 24 was reported.
Time Frame: At Week 24
Population: The SAF included all participants who received dupilumab.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 24
Percentage of Participants | 8.3 [1.03 to 27.00]

2. Secondary Outcome: Change From Baseline in Cumulative Tolerated Dose (Log Transformed) of Peanut Protein During a DBPCFC at Weeks 24 and 36
Description: Change from baseline in cumulative tolerated dose (log transformed) of peanut protein during a DBPCFC at Week 24 and Week 36 was reported.
Time Frame: Weeks 24 and 36
Population: The SAF included all participants who received dupilumab.
Measure: Mean (Standard Deviation); unit: Log Transformed Milligrams
Arm/Group | Dupilumab
Number analyzed (Participants) | 24
Log Transformed Milligrams
  Change at Week 24 | 0.69 (1.822)
  Change at Week 36: number analyzed (Participants) | 2
  Change at Week 36 | 3.38 (3.096)

3. Secondary Outcome: Percentage of Participants Treated With Dupilumab Who Passed a DBPCFC With at Least 444 mg (Cumulative) Peanut Protein at Week 36
Description: Symptoms considered to be allergic were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions. The scale is Grade 1 (Mild) through 5, the higher the grade, the more severe the allergic reaction. Participants were considered to have passed the DBPCFC if they did not experience any objective Grade 1 reaction. Only participants treated with dupilumab who passed at least 444 mg (cumulative) peanut challenge at Week 24 were eligible for Week 36 DBFC.
Time Frame: At Week 36
Population: A subset of the SAF that included only participants who passed the DBPCFC of at least 444 mg (cumulative) at Week 24.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 2
Percentage of Participants | 50.0

4. Secondary Outcome: Percentage of Participants Treated With Dupilumab Who Passed a DBPCFC With at Least 1044 mg (Cumulative) Peanut Protein at Week 24
Description: Symptoms considered to be allergic were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions. The scale is Grade 1 (Mild) through 5, the higher the grade, the more severe the allergic reaction. Participants were considered to have passed the DBPCFC if they did not experience any objective Grade 1 reaction. Percentage of participants treated with dupilumab who passed a DBPCFC with at least 1044 mg (cumulative) peanut protein at Week 24 was reported.
Time Frame: At Week 24
Population: The SAF included all participants who received dupilumab.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 24
Percentage of Participants | 0.0 [0.00 to 14.25]

5. Secondary Outcome: Percentage of Participants Treated With Dupilumab Who Passed a DBPCFC With at Least 1044 mg (Cumulative) Peanut Protein at Week 36
Description: as for outcome 3
Time Frame: At Week 36
Population: A subset of the SAF that included only participants who passed the DBPCFC of at least 444 mg (cumulative) at Week 24.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 2
Percentage of Participants | 50.0

6. Secondary Outcome: Percentage of Participants Treated With Dupilumab Who Passed a DBPCFC With at Least 2044 mg (Cumulative) Peanut Protein at Week 24
Description: Symptoms considered to be allergic were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions. The scale is Grade 1 (Mild) through 5, the higher the grade, the more severe the allergic reaction. Participants were considered to have passed the DBPCFC if they did not experience any objective Grade 1 reaction. Percentage of participants treated with dupilumab who passed a DBPCFC with at least 2044 mg (cumulative) peanut protein at Week 24 was reported.
Time Frame: At Week 24
Population: The SAF included all participants who received dupilumab.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 24
Percentage of Participants | 0.0 [0.00 to 14.25]

7. Secondary Outcome: Percentage of Participants Treated With Dupilumab Who Passed a DBPCFC With at Least 2044 mg (Cumulative) Peanut Protein at Week 36
Description: as for outcome 3
Time Frame: At Week 36
Population: A subset of the SAF that included only participants who passed the DBPCFC of at least 444 mg (cumulative) at Week 24.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 2
Percentage of Participants | 0.0

8. Secondary Outcome: Percent Change From Baseline in Peanut-specific Immunoglobulin E (sIgE) at Weeks 4, 8, 12, 16, 24, and 36
Description: Percent change from baseline in sIgE at Weeks 4, 8, 12, 16, 24, and 36 was reported.
Time Frame: Weeks 4, 8, 12, 16, 24, and 36
Population: The SAF included all participants who received dupilumab.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Dupilumab
Number analyzed (Participants) | 24
Percent Change
  Percent change at Week 4 | -7.86 [-19.75 to -1.62]
  Percent change at Week 8 | -21.03 [-33.45 to -10.37]
  Percent change at Week 12: number analyzed (Participants) | 23
  Percent change at Week 12 | -32.10 [-40.92 to -11.14]
  Percent change at Week 16 | -32.22 [-47.75 to -16.17]
  Percent change at Week 24 | -49.25 [-61.22 to -31.85]
  Percent change at Week 36 | -58.43 [-71.25 to -45.17]

9. Secondary Outcome: Change From Baseline in Titrated Skin Prick Test (SPT) Measured by Average Wheal Size Area Under the Curve (AUC) After Peanut Allergen Stimulation at Different Concentrations at Weeks 4, 12, 24, and 36
Description: The titrated SPT is the skin testing for atopic response at different concentrations of peanut extract with saline as negative control and histamine as positive controls. Wheal size induced by peanut extract at each concentration was calculated as average of largest diameter and perpendicular midpoint diameter. The AUC for titrated SPT was calculated using the mean wheal diameter versus the concentration at which the wheal diameter was measured, which was then normalized to concentration. Change from baseline in titrated SPT as measured by average wheal size AUC after peanut allergen stimulation at different concentrations at Weeks 4, 12, 24, and 36 was reported.
Time Frame: Weeks 4, 12, 24, and 36
Population: The SAF included all participants who received dupilumab.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Dupilumab
Number analyzed (Participants) | 24
millimeter (mm)
  Change at Week 4 | -0.633 (2.0604)
  Change at Week 12 | -0.174 (2.0618)
  Change at Week 24 | -0.232 (2.0610)
  Change at Week 36: number analyzed (Participants) | 23
  Change at Week 36 | -0.364 (2.1419)

10. Secondary Outcome: Percentage of Participants With Grade 2 or Above Allergic Reactions During the DBPCFC at Week 24
Description: Symptoms considered to be allergic were graded using the Consortium of Food Allergy Research (CoFAR) Grading Scale for Systemic Allergic Reactions. The scale is Grade 1 (Mild) through 5, the higher the grade, the more severe the allergic reaction. Percentage of participants with Grade 2 (Moderate) or above allergic reactions during the DBPCFC at Week 24 was reported.
Time Frame: At Week 24
Population: The SAF included all participants who received dupilumab.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 24
Percentage of Participants | 33.3

11. Secondary Outcome: Percentage of Participants Who Used Epinephrine as a Rescue Medication During the DBPCFC at Week 24
Description: Percentage of participants who used Epinephrine as a rescue medication during the DBPCFC at Week 24 was reported.
Time Frame: At Week 24
Population: The SAF included all participants who received dupilumab.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 24
Percentage of Participants | 41.7

ADVERSE EVENTS:
Time Frame: Up to the end of study (Week 36)
Arm/Group | Placebo | Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/24
Other Adverse Events (participants affected / at risk) | 0/1 | 11/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1) | Dupilumab (N=24)
Injection site erythema (General disorders) | 0 (0) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 2 (3)
Injection site pain (General disorders) | 0 (0) | 3 (4)
Injection site reaction (General disorders) | 0 (0) | 2 (4)
Injection site urticaria (General disorders) | 0 (0) | 3 (5)
Medical device pain (General disorders) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (8)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT03793608/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT03793608/SAP_002.pdf